CLINICAL TRIAL: NCT02195284
Title: An Open-label Study of Inhaler Device Attributes Investigating Critical and Overall Errors, and Ease of Use and Preference Between a Number of Inhaler Devices (ELLIPTA, DISKUS/ACCUHALER, TURBUHALER, and MDI) in Adult Subjects With Asthma (Study 200330)
Brief Title: To Study Device Attributes by Investigating Errors Made in Use, Ease of Use and Preference Among Different Inhalers in Subjects With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 200330
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-09

CONDITIONS: Asthma
Keywords: Inhaler preference; Overall inhaler error; DISKUS/ACCUHALER; MDI; TURBUHALER; ELLIPTA; Ease of use; Critical inhaler error
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sub-study 1 (Experimental): Subjects will be randomized to either use ELLIPTA inhaler first and then DISKUS/ACCUHALER inhaler or use DISKUS/ACCUHALER inhaler first and then ELLIPTA inhaler
  Interventions: Device: ELLIPTA; Device: DISKUS/ACCUHALER
- Sub-study 2 (Experimental): Subjects will be randomized to either use ELLIPTA inhaler first and then MDI (metered-dose inhaler) or use MDI first and then ELLIPTA inahler
  Interventions: Device: ELLIPTA; Device: MDI
- Sub-study 3 (Experimental): Subjects will be randomized to either use ELLIPTA inhaler first and then TURBUHALER inhaler or use TURBUHALER inhaler first and then ELLIPTA inhaler
  Interventions: Device: ELLIPTA; Device: TURBUHALER

INTERVENTIONS:
Device: ELLIPTA — Dry powder inhaler (placebo) with two blister strips. One placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate
Device: DISKUS/ACCUHALER — Placebo inhaler with one blister strip containing lactose monohydrate.
  Arms: Sub-study 1
Device: MDI — Placebo inhaler containing propellant (1,1,1, 2-Tetrafluoroethane)
  Arms: Sub-study 2
Device: TURBUHALER — Placebo inhaler containing lactose monohydrate.
  Arms: Sub-study 3

SUMMARY:
This study is designed to assess the proportion of asthma subjects making critical and non-critical errors made in using ELLIPTA® inhaler compared with other commercially available inhaler devices such as the TURBUHALER®, MDI (metered-dose inhaler), and DISKUS/ACCUHALER®. This study will also assess the ease of use and preference between the ELLIPTA inhaler and the other commercially available inhaler devices. This is a randomized, open-label, placebo, crossover, multicentre study with a single visit. The study will comprise three sub-studies. Subjects will receive inactive treatment (placebo) via the ELLIPTA inhaler and one of the other inhaler devices depending on the sub-study they are allocated to. Only subjects who are naïve to the ELLIPTA inhaler and to one of the other inhalers that will be used in this study will be included. The study will be conducted in the Netherlands and the UK, and comprises one visit only. A sufficient number of subjects (at least 190) with asthma will be screened and 180 will be randomized to one of the three sub-studies. Eligible subjects will be allocated to one of the sub-studies in the following order depending on their experience of using the other inhaler (i.e., depending on which other inhaler they are naïve to).

ELLIPTA, DISKUS, and ACCUHALER are registered trademarks of the GSK group of companies. TURBUHALER is a registered trademark of AstraZeneca.

DETAILED DESCRIPTION:
This is a non-interventional study and not an observational study and therefore some fields are not applicable for the CT.gov observational study design. It would be preferential to have the field populated as "not applicable" for sampling method, time perspective, and observational study model as they don't apply to this study design.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: Subject must give their signed and dated written informed consent to participate; Subject understands and is willing, able, and likely to comply with study procedures and restrictions; Subject must be able to read, comprehend, and record information in Dutch and/or English
* Age: >=18 years of age
* Gender: Male or female subjects.
* Asthma Diagnosis: A diagnosis of asthma as defined by the National Institutes of Health. Comorbidities (rheumatoid arthritis or other locomotor problems, visual impairment, and depression or anxiety) will be documented as relevant to inhaler use.
* Asthma treatment: All subjects should be currently receiving treatment for asthma.
* Must be naive to using ELLIPTA inhaler and at least one other inhaler device.

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease (COPD): Subjects with a current diagnosis of COPD only.
* Contraindications: A history of allergy or hypersensitivity to lactose/milk protein or magnesium stearate or to any other excipient.
* Subjects who are currently participating in another randomised pharmacological interventional trial.
* Inability to Read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a questionnaire and understand verbal instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects making at least one critical error after reading the patient information leaflet | Day 1
  In each sub-study, subjects will be asked to read the patient instruction leaflet of the first device and then asked to demonstrate inhaler use. Any errors (critical or non-critical) made by the subject while using the first inhaler will be recorded by the health care professional (HCP). The same procedures will be followed for the second inhaler. A critical error is defined as an error that is most likely to result in no or only minimal medication being inhaled

SECONDARY OUTCOMES:
Percentage of subjects making at least one critical error after the first instruction from HCP | Day 1
  In each sub-study, if the subject makes any error while demonstrating the use of the first inhaler after reading the patient instruction leaflet, the HCP will demonstrate the correct use of the inhaler to the subject. The subject will then be asked to demonstrate inhaler use again. Any errors will be recorded by the HCP. The same procedures will be followed for the second inhaler. A critical error is defined as an error that is most likely to result in no or only minimal medication being inhaled
Percentage of subjects making at least one overall error after reading the patient information leaflet | Day 1
  In each sub-study, subjects will be asked to read the patient instruction leaflet of the first device and then asked to demonstrate inhaler use. Any errors (critical or non-critical) made by the subject while using the first inhaler will be recorded by the HCP. The same procedures will be followed for the second inhaler. An overall error includes a critical and non-critical error
The percentage of subjects making at least one overall error after the first instruction on use by the HCP | Day 1
  In each sub-study, if the subject makes any error while demonstrating the use of the first inhaler after reading the patient instruction leaflet, the HCP will demonstrate the correct use of the inhaler to the subject. The subject will then be asked to demonstrate inhaler use again. Any errors (critical or non-critical) will be recorded by the HCP. The same procedures will be followed for the second inhaler. An overall error includes a critical and non-critical error
The number of instructions (maximum three times) from the HCP which are needed to demonstrate adequate inhalation technique | Day 1
  In each sub-study, if the subject makes any error while demonstrating the use of the first inhaler after reading the patient instruction leaflet, the HCP will demonstrate the correct usage of the inhaler to the subject. The subject will then be asked to demonstrate inhaler use again. Any errors will be recorded by the HCP. The same procedures will be repeated if the subject continues to make errors in the use of the inhaler. In total, the HCP will demonstrate the use of the inhaler up to three times. Same procedures will be followed for second inhaler.
The percentage of subjects who prefer the ELLIPTA device compared to the other devices as assessed by the 'preference' questionnaire | Day 1
  After completing the demonstration procedures of the inhalers, the HCP will ask the subject a number of questions from preference questionnaire after completing the ease of use questionnaire. Preference questionnaire will consist of eight questions with each question having one response to chose from 3 options of preference (Other inhaler device, ELLIPTA inhaler device, No preference)
The percentage of subjects who found the ELLIPTA device 'easy to use' compared with the other devices' as assessed by the 'ease of use' questionnaire | Day 1
  After completing the demonstration procedures of the inhalers, the HCP will ask the subject a number of questions from ease of use questionnaire. Ease of use questionnaire will consist of six questions each for ELLIPTA inhaler and the other inhaler under study. Each question will have one response to chose from 5 options of ease of use (Very easy, easy, neutral, difficult and very difficult)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Netherlands (2):
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Zutphen
- United Kingdom (2):
  - GSK Investigational Site, Portsmouth
  - GSK Investigational Site, Southampton

REFERENCES:
- [Derived] van der Palen J, Thomas M, Chrystyn H, Sharma RK, van der Valk PD, Goosens M, Wilkinson T, Stonham C, Chauhan AJ, Imber V, Zhu CQ, Svedsater H, Barnes NC. A randomised open-label cross-over study of inhaler errors, preference and time to achieve correct inhaler use in patients with COPD or asthma: comparison of ELLIPTA with other inhaler devices. NPJ Prim Care Respir Med. 2016 Nov 24;26:16079. doi: 10.1038/npjpcrm.2016.79. PMID 27883002